CLINICAL TRIAL: NCT02012608
Title: Glutamine for the Prevention of Radiation Toxicity in Subjects Undergoing Breast Conserving Therapy
Brief Title: Glutamine for the Prevention of Radiation Toxicity in Subjects Conserving Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding/ PI leaving institution
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202253
Record Dates: First submitted 2013-12-03; First posted 2013-12-16 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Glutamine; Glucose; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine (Active Comparator): Powdered Glutamine, 10.0 grams by mouth three times a day (TID) for 30 days, so that daily dose is 30 grams per day
  Interventions: Drug: Glutamine
- Placebo (Placebo Comparator): Powdered Dextrose, 8.33 grams by mouth TID for 30 days, so that daily dose is 25 grams per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glutamine — Oral glutamine for subjects undergoing breast conserving therapy
  Other Names: Gln; Q
  Arms: Glutamine
Drug: Placebo — For subjects undergoing breast conserving therapy
  Other Names: Dextrose; Dextrose monohydrate; Sugar
  Arms: Placebo

SUMMARY:
This study is a single-centered, double-blind, two-arm randomized study to determine if oral glutamine will reduce radiation toxicity for the subjects undergoing Breast Conserving Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject have been diagnosed with Stage I or II invasive breast cancer
* Subject will undergo Accelerated Partial Breast Irradiation (APBI) as part of Breast Conserving Therapy (BCT)
* Subject is eligible for APBI based on American Society of Therapeutic Radiation Oncology (ASTRO) criteria
* Subject is 18 years of age or older
* Subject is female

Exclusion Criteria:

* History of uncontrolled, clinically significant lung, heart, endocrine, liver, or renal disease
* Subject has been diagnosed with any other cancer
* Subject has a known hypersensitivity reaction to the following: oral glutamine (GLN), glutamate, monosodium glutamate (MSG) (i.e., Chinese restaurant syndrome)
* Subject has history of collagen vascular disease
* Subject has been diagnosed with Diabetes mellitus I or II
* Subject has had any prior breast radiation
* Subject is pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loverd Peacock, MD, Principal Investigator — University of Arkansas; Yihong Kaufmann, PhD, Study Chair — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glutamine | Placebo
Started | 7 | 7
Completed | 4 | 7
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Excessive Radiation Toxicity as Defined by Radiation Therapy Oncology Group (RTOG) Acute Scale of Radiation-toxicity Criteria
Description: The primary efficacy outcome will be excessive toxicity, which will be defined as a score of 2 or higher using the Radiation Therapy Oncology Group (RTOG) Acute scale of radiation-toxicity criteria when scored on either the 12-day or 30-day assessment time.
  The RTOG scale ranges from 0-4 with 0 being defined as "no change".
Time Frame: 12 days and 30 days
Population: No data displayed because Outcome Measure has zero total participants analyzed and no data was collected.
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Glutamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutamine (N=7) | Placebo (N=7)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
skin erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 2 (2) | 0 (0)
asymptomatic breast edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
breast fibrosis/fat necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
decreased lymphocyte count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
increased alkaline phosphatase (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
chloride out of range (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Outcome measures not computed because data would not be statistically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02012608/Prot_SAP_000.pdf